CLINICAL TRIAL: NCT03361202
Title: Evolution of Microparticles Circulating Plasma Concentration in Atrial Fibrillation After Percutaneous Occluding of the Left Atrium With Prosthesis (Amplatzer® Cardiac Plug)
Brief Title: Microparticles Circulating Plasma Concentration in Atrial Fibrillation After Percutaneous Occluding of the Left Atrium
Acronym: MICROPLUG
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Institut Mutualiste Montsouris (Other)
Collaborators: Société Française de Cardiologie (Other)
Responsible Party: Sponsor
Other Study IDs: CARDIO-01-2015
Record Dates: First submitted 2016-09-12; First posted 2017-12-04 (Actual); Last update posted 2017-12-04 (Actual); Status verified 2017-09

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — 4 ml of arterial or venous blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Atrial fibrillation group: blood sampling
  Interventions: Other: blood sampling
- control group: blood sampling
  Interventions: Other: blood sampling

INTERVENTIONS:
Other: blood sampling — * atrial fibrillation group:before Percutaneous Occluding of the Left Atrium, at hospital discharge and at J45 follow up
  * control group:before coronary angiography and at hospital discharge.

SUMMARY:
The aim of the study is to compare levels of differnts types of microparticles circulating before and after percutaneous occluding of the left atrium by patients with atrial fibrillation and patients control.

Hypothesis is that prothesis implantation will decrease levels of microparticles circulating in blood circulation because of occluding of the left atrium .

ELIGIBILITY:
Inclusion Criteria:

atrial fibrillation group:

* high embolic risk (CHADS-VASC2 score ≥4)
* formal and final contraindication to anticoagulant therapy
* no heart thrombus on ETO and TDM before percuraneous occluding

control group:

* suspicion of stable coronary artery disease, coronary angiography scheduled and double platelet aggregation (clopidogrel and aspirine)

Exclusion Criteria: for both groups

* congestive heart failure, severe aortic stenosis, EP or TVP early.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: two groups of patients:
  * control
  * atrial fibrillation
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2015-01 (Actual); Primary Completion 2018-01 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
levels of microparticles expressing phosphatidylserine in atrial fibrillation group | 45 days after Percutaneous Occluding of the Left Atrium.
  blood samples analized by flow cytometry

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas AMABILE, Principal Investigator — Institut Mutualiste Montsouris
Locations (1):
- Institut Mutualiste Montsouris, Paris, France

IPD SHARING:
Plan to Share IPD: No